CLINICAL TRIAL: NCT06814483
Title: Modulation Effects of a Computer-based Multimodal Mind and Body Approach for Mild Cognitive Decline
Brief Title: Effects Multimodal Mind and Body Approach for MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Principal investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022p003426
Record Dates: First submitted 2025-01-27; First posted 2025-02-07 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment
Keywords: mind-body intervention; Baduanjin; Cognitive training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A computer-based multimodal mind and body approach (cbMMBA) (Experimental): cbMMBA will include three modules: BDJ (module 1), acupressure (module 2), and relaxation techniques including deep breathing, guided imagery, and progressive muscle relaxation
  Interventions: Behavioral: Experimental: A computer-based multimodal mind and body approach (cbMMBA)
- a standard cognitive training (Active Comparator): The program uses paper puzzles (Sudoku, crosswords, word-search, etc.) to engage subjects
  Interventions: Behavioral: A standard cognitive training group

INTERVENTIONS:
Behavioral: Experimental: A computer-based multimodal mind and body approach (cbMMBA) — cbMMBA will include three modules: BDJ, acupressure, and relaxation techniques including deep breathing, guided imagery, and progressive muscle relaxation.
  Arms: A computer-based multimodal mind and body approach (cbMMBA)
Behavioral: A standard cognitive training group — The program uses paper puzzles (Sudoku, crosswords, word-search, etc.) to engage subjects
  Arms: a standard cognitive training

SUMMARY:
The aim of this application is to develop a computer-based multimodal mind and body approach (CMMBA) for mild cognitive impairment (MCI). This product will provide a new, cost-effective and easily accessible treatment option for MCI and potentially other age-related dementia.

DETAILED DESCRIPTION:
The goal of this Phase I R41 (STTR) application is to develop a computer-based multimodal mind and body approach (cbMMBA) to improve the cognitive function for mild cognitive impairment (MCI). This application, if successful, will provide a cost-effective and easily accessible treatment option for MCI and other age-related dementia, significantly improve the prevention of MCI development, and directly benefit patients suffering from the highly prevalent disorder, particularly for those who may have limited access to in-person mind and body interventions.

ELIGIBILITY:
Inclusion Criteria:

1. report of cognitive decline / complaint by the patient, the patient's informant, or the physician;
2. cognitive impairment is confirmed by objective cognitive measures (Montreal Cognitive Assessment (MoCA) and neuropsychological testing), where objective cognitive impairment is defined as poor performance in one or more cognitive measures suggesting deficit in one or more cognitive domains;
3. patient has preserved independence in functional abilities (measured by informant report, completion of Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) checklists);
4. not demented;

Exclusion Criteria:

1. has severe visual or hearing impairment;
2. has pre-existing musculoskeletal or other conditions, which prohibit BDJ performance and / or the application of acupressure at the selected points;
3. has suffered from a neurological disorder (e.g., severe head trauma), psychiatric disease (e.g., major depression), or any other major medical disease that could potentially compromise their cognition;
4. has had prior experience with BDJ or acupressure or relaxation techniques in the past year.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
The Small Business Act permits SBIR/STTR grantees to withhold data for 4 years after the end of the grant award.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A Computer-based Multimodal Mind and Body Approach (cbMMBA) | a Standard Cognitive Training
Started | 17 | 15
Completed | 11 | 15
Not Completed | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Computer-based Multimodal Mind and Body Approach (cbMMBA) | a Standard Cognitive Training | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Continuous [Mean (Standard Deviation); unit: year] | 73.06 (9.91) | 72.73 (7.36) | 72.91 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Proportion of subjects who complete all assessments from the total number of subjects started the first intervention
Time Frame: Through study intervention, an average of three months
Measure: Count of Participants; unit: Participants
Arm/Group | A Computer-based Multimodal Mind and Body Approach (cbMMBA) | a Standard Cognitive Training
Number analyzed (Participants) | 14 | 15
Participants | 11 | 15

2. Primary Outcome: Fidelity
Description: session completed of total 30 classes
Time Frame: Through study interventions, an average of three months
Measure: Mean (Standard Deviation); unit: session
Arm/Group | A Computer-based Multimodal Mind and Body Approach (cbMMBA) | a Standard Cognitive Training
Number analyzed (Participants) | 17 | 15
session | 25.6 (7.9) | 29.5 (1.1)

3. Primary Outcome: Satisfaction to Intervention
Description: average score in a 1-5 scale, 5 indicates very satisfied with the intervention
Time Frame: Through study interventions, an average of three months
Measure: Mean (Standard Deviation); unit: points in a 1-5 scale
Arm/Group | A Computer-based Multimodal Mind and Body Approach (cbMMBA) | a Standard Cognitive Training
Number analyzed (Participants) | 14 | 15
points in a 1-5 scale | 4.8 (0.42) | 4.5 (0.64)

4. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events were assessed by participant self-report at each study visit. An adverse event was defined as any unfavorable or unintended sign, symptom, or medical occurrence temporally associated with study participation, regardless of attribution. This outcome reports the number of participants who experienced ≥1 adverse event during the study period (each participant counted once).
Time Frame: Through study interventions, an average of three months
Measure: Count of Participants; unit: Participants
Arm/Group | A Computer-based Multimodal Mind and Body Approach (cbMMBA) | a Standard Cognitive Training
Number analyzed (Participants) | 17 | 15
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 6 month
Arm/Group | A Computer-based Multimodal Mind and Body Approach (cbMMBA) | a Standard Cognitive Training
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 2/17 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A Computer-based Multimodal Mind and Body Approach (cbMMBA) (N=17) | a Standard Cognitive Training (N=15)
planned heart surgery (Cardiac disorders) | 1 (1) | 0 (0) — unrelated to intervention
PTSD recurrence (Psychiatric disorders) | 1 (1) | 0 (0) — unrelated to the intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT06814483/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT06814483/SAP_001.pdf